CLINICAL TRIAL: NCT05702073
Title: A Randomized, Open-Label, Controlled, Parallel-group, Multicenter Trial Comparing the Efficacy and Safety of INS068 and Insulin Glargine in Subjects With Type 2 Diabetes Mellitus Not Adequately Controlled With Basal Insulin
Brief Title: To Compare the Efficacy and Safety of INS068 and Insulin Glargine in Subjects With Type 2 Diabetes Mellitus Treated With Basal Insulin.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS068-301
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Controlled, Parallel-group, Multicenter Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INS068 (Experimental)
  Interventions: Drug: INS068 injection
- IGlar (Active Comparator)
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: INS068 injection — INS068 injected subcutaneously once daily. Treat-to-target dose titration during the trial
  Arms: INS068
Drug: Insulin Glargine — Insulin Glargine injected subcutaneously once daily. Treat-to-target dose titration during the trial
  Arms: IGlar

SUMMARY:
The study aims to evaluate the efficacy and safety of INS068 once daily (QD) in subjects with type 2 diabetes not adequately controlled with basal insulin compared to insulin Glargine QD for 26weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes≥ 6 months;
2. HbA1c 7.0% ~ 10.0% (Both inclusive) at screening;
3. Treated with Basal insulin ≥10U /day for at least 8 weeks prior to screening.

Exclusion Criteria:

1. Known or suspected allergy or intolerance to investigational medicinal products or related products.
2. Hospitalization for diabetic ketoacidosis or hyperglycemic hyperosmolar state within the previous 6 months.
3. Potentially unstable diabetic retinopathy or macular degeneration that requires treatment (e.g., laser, surgical, or injectable medications) within the previous 6 months.
4. Received premixed insulin, mealtime insulin, or insulin pump therapy within 8 weeks prior to screening.
5. Participated in clinical trials of any approved or unapproved investigational drug/treatment within the previous 1 month or 5 half-life period, whichever is longer, prior to screening.
6. Women who are pregnant, breastfeeding or planning to conceive, or women of childbearing potential are reluctant to use appropriate contraception during the trial and for at least 14 days after the last dose of the investigational medicinal drug; Anycircumstances that the investigator judges might not be suitable to participate in the trial..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0 to Week 26
  Change from baseline in Glycosylated Haemoglobin after 26 weeks of treatment

SECONDARY OUTCOMES:
Change in FPG(fasting plasma glucose) | Week 0 to Week 26
  Change from baseline in FPG after 26 weeks of treatment
Proportion of Subjects with HbA1c<7% and HbA1c≤6.5% | Week 0 to Week 26
  Proportion of subjects with HbA1c<7% and HbA1c≤6.5% after 26 weeks of treatment
per-breakfast SMPG | Week 0 to Week 26
  Mean and Within-subject variability of pre-breakfast SMPG after 26 weeks of treatment
8-point SMPG profiles | Week 0 to Week 26
Average daily Insulin dose | Week 0 to Week 26
  Average daily Insulin dose after 26 weeks of treatment.
Proportion of Subjects requiring rescue therapy during treatment | Week 0 to Week 26
  Proportion of subejcts requiring rescue therapy during 26 weeks of treatment
Frequency and severity of adverse events | Week 0 to Week26 +14 days follow-up
  Severity (mild, moderate and severe) is assessed by investigator.
Incidence and rate of Hypoglycemic events | Week 0 to Week 26+14 days follow-up
  Incidence and rate of of Hypoglycemic events
Change in weight | Week 0 to Week 26
  Change from baseline in weight after 26weeks of treatment
Anti-drug Antibodies | Week 0 to Week26 + 14 days follow-up
  Number of subjects with Positive Anti-drug Antibodies
Serum INS068 concentration | Week 0 to Week 26
  To evaluate PK of INS068
Change in scores of diabetes treatment satisfaction questionnaire status version (DTSQs) | Week 0 to Week 26
  Change from baseline in scores of DTSQs after 26 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided